CLINICAL TRIAL: NCT06614166
Title: Food Trial to Evaluate the Kinetics of the Medical Foods SBD111 and SBD121 Persistence in Healthy Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Solarea Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00078728
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Product Persistence in GI Tract; Kinetics; Rheumatoid Arthritis (RA); Bone Density
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Synbiotic Medical Food SBD111 (Experimental): Probiotic comprised of three lactic acid bacteria and one yeast
  Interventions: Other: SBD111 Probiotic Medical Food
- Synbiotic Medical Food SBD121 (Experimental): Probiotic comprised of three lactic acid bacteria and one bacillus
  Interventions: Other: SBD121 Probiotic Medical Food

INTERVENTIONS:
Other: SBD111 Probiotic Medical Food — Medical food comprised of probiotics and prebiotic fibers
  Arms: Synbiotic Medical Food SBD111
Other: SBD121 Probiotic Medical Food — Probiotic medical food comprised of three lactic acid bacteria and one bacillus
  Arms: Synbiotic Medical Food SBD121

SUMMARY:
This study is a randomized, open-label, trial in healthy volunteers. Trial participants will be given a medical food product (combination of probiotics and prebiotics) called SBD111 or SBD121 for seven days and microbial abundance in feces will be measured during that time and for four weeks following administration.

DETAILED DESCRIPTION:
This DMA persistence food trial provides critical complimentary data to the ongoing efficacy food trials of SBD111 and SBD121 medical foods. While the SBD111 and SBD121 medical food products have been tested in multiple preclinical studies, GLP-Toxicity studies in Rats, and ongoing safety and efficacy trials, no study has yet examined how quickly these DMAs become detectable/active in human stool samples or the rate they clear from human stool following treatment cessation. The data provided by this study could inform the interpretation efficacy trial data with regard to subject adherence.

Objectives The primary goal of this study is to evaluate the prevalence and persistence of SBD111 and SBD121 medical foods, two novel combinations of probiotics and prebiotic dietary fibers, over time in stool samples. We will determine the effect of these Defined Microbial Assemblages (DMAs) on fecal microbiota composition and functional potential, as well as the duration of SBD111 and SBD121 product persistence in the gastrointestinal tract. DMAs will be administered for 7 days, and stool samples will be collected during DMA administration and up to 28 days post DMA cessation for microbial DNA extraction. Fecal microbial DNA will be subjected to qPCR and high throughput shotgun sequencing to determine the presence and amount of DMA microbes that are present before, during, and after DMA administration. We will also use the resulting shotgun sequencing data to determine whether any taxonomic shifts or functional changes occur in response to DMA administration and/or cessation. Finally, as an exploratory measure, we will attempt to isolate live DMA microbes from participants' fecal samples using microbiological techniques.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Stated availability throughout entire study period and willingness to fulfill all details of the protocol.
3. Age 18-64 years.
4. Be in general good health as determined by a screening evaluation within 30 days of the first dose of SBD111 or SBD121.
5. Willing to comply with protocol and report on compliance and side effects during study period.
6. Body Mass Index between 18.5 and 35 kg/m2.

Exclusion Criteria:

1. Are currently taking probiotic or prebiotic supplements or have taken them in the past 30 days.
2. Unwilling to avoid probiotics/prebiotics supplements for the duration of the study.
3. Known or suspected allergies to probiotics, maltodextrin, or berries.
4. Received oral or parenteral antibiotics within 3 months of enrollment or prescribed antibiotics on the day of enrollment.
5. Major surgery on the intestines or endoscopy within last 3 months.
6. Current smoker.
7. History of drug and/or alcohol abuse at the time of enrollment.
8. Presence of any of the following:
9. Abnormal vital signs or clinically significant systems abnormalities based on screening questionnaire.
10. Indwelling catheter or implanted hardware/prosthetic device or feeding tube.

    a. Excluding joint replacements
11. Febrile illness (oral temperature >37 degrees Celsius) or one or more episodes of diarrhea within 72 hours of baseline (first dose of study article).
12. Active bowel leak, acute abdomen, colitis, or active GI disease or history of gastric or intestinal dysmotility, slowed transit time, variable small intestinal permeability, pancreatitis, or inflammatory bowel disease.
13. History of Hepatitis B or Hepatitis C infections, cirrhosis, or chronic liver disease.
14. Underlying structural heart disease or previous history of endocarditis or valve replacement.
15. Immunosuppression including HIV positive, solid organ or stem cell transplant recipient, receiving any oral or parenteral immunosuppressive therapy.
16. History of Celiac disease.
17. History of cancer.
18. Excluding non-melanoma skin cancers or cancer more than 10 years ago.
19. History of autoimmune disease and taking any immunosuppressant drugs.
20. Active TB.
21. Women only - pregnant, planning on becoming pregnant within the next 2 months, breastfeeding, positive urine pregnancy test within 24 hours of first dose of DMA.
22. Participants may be excluded if, in the investigator's opinion, there is evidence of cognitive impairment or dementia which is sufficient to interfere with informed consent or adherence to the study protocol. Four questions will be asked during the informed consent process to confirm participant's understanding and ability to comply.
23. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer participating in the study or would make it unlikely the volunteer could complete the study.
24. Bowel movement frequency less than one per 36-hour period.
25. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-05-23 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Persistence of SBD111 and SBD121 microbes in fecal samples | 5 weeks
  DNA isolated from fecal swabs will be used to determine the persistence of SBD111 and SBD121 microbes in stool samples up to 28 days following twice-daily oral administration of SBD111 or SBD121 to healthy adults.

SECONDARY OUTCOMES:
Microbial Community Structure Changes | 5 weeks
  Using metagenomic sequencing, we will assess microbial community structural and functional changes that occur during and up to 28 days following twice-daily oral administration of SBD111 or SBD121 to healthy adults. This will be done via sequence assessment of microbiota taxonomies and functional genes.

OTHER OUTCOMES:
Microbe Viability | 2 weeks
  From frozen fecal samples we will assess the viability of SBD111 and SBD121 microbes in fecal samples after 0, 7, and 14 days of oral administration using standard microbiological plating techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia E Ballok, PhD, Principal Investigator — Solarea Bio, Inc
Locations (1):
- Solarea Bio Inc, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- [Background] Easson DD Jr, Murphy VA, Ballok AE, Soto-Giron MJ, Miller KJ, Charbonneau MR, Schott EM, Greene T, Rodricks J, Toledo GV. Food safety assessment and 28-day toxicity study of the synbiotic medical food consortium SBD121. Food Chem Toxicol. 2024 Sep;191:114839. doi: 10.1016/j.fct.2024.114839. Epub 2024 Jun 26. PMID 38942165
- [Background] Easson DD Jr, Murphy VA, Ballok AE, Soto-Giron MJ, Schott EM, Rodricks J, Toledo GV. Food safety assessment and toxicity study of the synbiotic consortium SBD111. Food Chem Toxicol. 2022 Oct;168:113329. doi: 10.1016/j.fct.2022.113329. Epub 2022 Aug 7. PMID 35948142
- [Background] Lawenius L, Gustafsson KL, Wu J, Nilsson KH, Moverare-Skrtic S, Schott EM, Soto-Giron MJ, Toledo GV, Sjogren K, Ohlsson C. Development of a synbiotic that protects against ovariectomy-induced trabecular bone loss. Am J Physiol Endocrinol Metab. 2022 Apr 1;322(4):E344-E354. doi: 10.1152/ajpendo.00366.2021. Epub 2022 Feb 14. PMID 35156423